CLINICAL TRIAL: NCT01097902
Title: Experimental Inflammatory and Micro-incisional Pain Model Analysis by Gene Expression and Interstitial Fluid Proteomics of Skin Tissue
Brief Title: Study of Experimental Models of Pain and Inflammation.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Martin Angst (Other)
Responsible Party: Sponsor-Investigator, Martin Angst, Professor of Anesthesia, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: SU-03012010-5102
Record Dates: First submitted 2010-03-31; First posted 2010-04-02 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Pain; Inflammation
MeSH Terms: conditions — Pain; Inflammation | interventions — Ibuprofen; Drugs, Generic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Ibuprophen 800 mg (Active Comparator): Oral ibuprofen 800 mg, administered 24 hours after exposure to UV radiation for the creation of an inflamed lesion, and 2 hours prior to site evaluation.
  Interventions: Drug: Ibuprofen
- Placebo (Placebo Comparator): Oral placebo administered 24 hours after exposure to UV radiation for the creation of an inflamed lesion, and 2 hours prior to site evaluation.
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: Ibuprofen — 800 mg oral one time only
  Other Names: Ibuprofen, generic
  Arms: Ibuprophen 800 mg
Drug: Placebo tablet — Placebo tablet oral one time only
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The experimental pain model studied in this proposal show characteristics of an inflamed wound with a pro-inflammatory response. This study will help discover candidate genetic and/or proteomic pain biomarkers that could provide objective and mechanism based tests to diagnose, monitor or quantify pain. We also hope to determine the measurable effects of a known non-steroidal anti-inflammatory drug (NSAID) on biomarkers of pain and inflammation.

ELIGIBILITY:
Inclusion Criteria:1) Age 18-60 2) Skin type II or III according to classification of Fitzpatrick 3) Negative pregnancy test (women of childbearing potential) 4) Willing and able to sign an informed consent form and Health Insurance Portability and Accountability Act (HIPAA) authorization and to comply with study procedures

Exclusion Criteria:1) History of acute or chronic illness that may hinder study procedures or confuse interpretation of the data (e.g. dermatological, neurological, psychiatric or addictive diseases) 2) Clinically significant cardiovascular, pulmonary, hepatic or renal diseases 3) Major bodily injury within 3 months of study participation 4) Surgery within 3 months of study participation 5) Pregnancy or breast-feeding 6) Intake of prescription drugs with anti/pro-inflammatory action 7) Intake of prescription drugs with anti/pro-analgesic action 8) Inability to abstain from any anti/pro inflammatory drugs during the 24-hour period preceding a study session 9) Inability to abstain from any anti/pro-analgesic drugs during the 24-hour period preceding a study session 10) Prior medical history that would contraindicate the use of NSAID, or previous negative reaction to NSAIDs or aspirin 11) Inability to obtain at least 6 hours of sleep during the night preceding a study session

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Mechanical and thermal pain measurements, inflammatory COX and Prostaglandin E2 (PGE2) gene expression. | 48 hours

SECONDARY OUTCOMES:
Interleukin-1beta and Interleukin-8 regulation | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Martin S Angst, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] Angst MS, Clark JD, Carvalho B, Tingle M, Schmelz M, Yeomans DC. Cytokine profile in human skin in response to experimental inflammation, noxious stimulation, and administration of a COX-inhibitor: a microdialysis study. Pain. 2008 Sep 30;139(1):15-27. doi: 10.1016/j.pain.2008.02.028. Epub 2008 Apr 8. PMID 18396374
- [Background] Angst MS, Tingle M, Schmelz M, Carvalho B, Yeomans DC. Human in-vivo bioassay for the tissue-specific measurement of nociceptive and inflammatory mediators. J Vis Exp. 2008 Dec 1;(22):1074. doi: 10.3791/1074. PMID 19229167